CLINICAL TRIAL: NCT03451695
Title: Effect of Intrathecal Morphine on Chronic Pain After Elective Caesarean Section: A Randomized Controlled Trial.
Brief Title: Effect of Intrathecal Morphine on Chronic Pain After Elective Caesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Dr Asish Subedi, Doctor, B.P. Koirala Institute of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRC/1183/017
Record Dates: First submitted 2018-02-20; First posted 2018-03-02 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Chronic Pain Post-Procedural
MeSH Terms: interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morphine group (Experimental): Morphine group will receive intrathecal 11 mg of hyperbaric bupivacaine (2.2 mL 0.5%), 10 μg of fentanyl (0.2 ml) and 100 μg of preservative free morphine (0.1 ml).
  Interventions: Drug: Morphine
- Placebo group (Placebo Comparator): Placebo group will receive intrathecal 11 mg of hyperbaric bupivacaine (2.2 mL 0.5%), 10 μg of fentanyl (0.2 ml) and normal saline (0.1 ml).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Morphine — Morphine group will receive intrathecal 11 mg of hyperbaric bupivacaine (2.2 mL 0.5%), 10 μg of fentanyl (0.2 ml) and 100 μg of preservative free morphine (0.1 ml).
  Arms: Morphine group
Drug: Placebo — Placebo group will receive 11 mg of hyperbaric bupivacaine (2.2 mL 0.5%), 10 μg of fentanyl (0.2 ml) and normal saline (0.1ml)
  Arms: Placebo group

SUMMARY:
The incidence of chronic post-surgical pain (CPSP) after caesarean section (CS) is reported to be as high as 18%, reflecting it to be a significant clinical problem. Studies related to prevention of progression of acute post-CS pain to its chronicity are sparse. Current guidelines on post-CS analgesia recommend the use of intrathecal (IT) opioids to spinal anaesthesia for improved post-CS pain relief. Despite its frequent use, studies related to the IT morphine use and its association with post-CS chronic pain are lacking.

A recent prospective observation study revealed a significant reduction in persistent pain after CS when IT morphine was used as an adjuvant to spinal anaesthesia. However, there is no any randomized controlled trial (RCT) that has explored this association to date. We hypothesized that spinal morphine would reduce the incidence of persistent pain after CS.

DETAILED DESCRIPTION:
This prospective, randomised, double-blind trial will take place at B.P Koirala Institute of Health Sciences, a University hospital situated in Nepal. Approval for the study has been obtained from the institution ethical committee. After the trial is registered, recruitment of the patient will be initiated. Consent for the participation in the study will be obtained during pre-anaesthetic assessment visits in the evening before surgery. During this visit, preoperative anxiety level (hospital anxiety and depression scale), pain catastrophizing (assessed with pain catastrophizing scale), preoperative pain sensitivity (assessed with pain pressure threshold and tolerance) will be recorded. The investigator will also educate the patients regarding the use of NRS scores for postoperative pain and satisfaction ratings.

Patients will be randomly assigned in a 1:1 ratio to one of the two groups (morphine and placebo groups). Randomization will be done in variable block sizes (4/6/8) by an internet based random-number generator list.

Morphine group will receive intrathecal 11 mg of hyperbaric bupivacaine (2.2 mL 0.5%), 10μg of fentanyl (0.2 ml) and 100 μg of preservative free morphine (0.1 ml). Placebo group will receive 11 mg of hyperbaric bupivacaine (2.2 mL 0.5%), 10μg of fentanyl (0.2 ml) and normal saline (0.1ml).

Postoperatively, pain, opioid consumption, sedation, nausea or vomiting, pruritus, and respiratory depression in the postanesthesia care unit (time 0 hours) and at 2, 6, 12, 24, and 48 hours will be evaluated. The area of hyperalgesia around the surgical incision will be assessed at 48 hrs postoperatively using a von Frey filament.

Patient satisfaction from postoperative analgesia will be assessed using a 5-point scale (1 = very unsatisfied, 2 = unsatisfied, 3 = fair, 4 = satisfied and 5 = very satisfied). At 8 wks patients will be assessed for post-natal depression using Edinburgh postnatal depression scale.

Patients will be contacted by telephone by one of the blinded investigator at 3, 6 months after the surgery. The short form brief pain inventory will be used to determine post-CS chronic pain

ELIGIBILITY:
Inclusion Criteria:

* Woman in American Society of Anesthesiologists (ASA) physical status classification II with full-term singleton pregnancy undergoing planned CS under spinal anesthesia.

Exclusion Criteria:

* contraindication to spinal anaesthesia, height<150 cm, ASA > II, BMI> 40, allergy to any drug used in the study, recent opioid exposure, substance abuse, significant cardiovascular, renal, or hepatic disease; and known fetal abnormalities.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 290 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-12-26 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with the incidence of post surgery chronic pain at 3 months following elective caesarean section | 3 months after elective caesarean section
  To find the number of participants with the incidence of post surgery chronic pain at 3 months following elective caesarean section in those receiving Intrathecal morphine and normal saline

SECONDARY OUTCOMES:
Number of participants with the incidence of post surgery chronic pain at 6 months following elective caesarean section | 6 month after elective caesarean section
  To find the number of participants with the incidence of post surgery chronic pain at 6 months following elective caesarean section in those receiving Intrathecal morphine and normal saline
Brief pain inventory (BPI) pain severity scores at 3 and 6 month after elective caesarean section between those receiving intrathecal morphine and normal saline | 3 and 6 months after elective caesarean section
  Short form Brief pain inventory (BPI) pain severity scores: Pain is rated on a 0 to 10 numerical rating scale, with 0="no pain" or and 10=pain "as bad as you can imagine." Participants rate their worst, least, and average pain over the last seven days, as well as their pain right now.
Brief Pain Inventory (BPI) pain interference scores at 3 and 6 month after elective caesarean section between those receiving intrathecal morphine and normal saline | 3 and 6 months after elective caesarean section
  Short form Brief pain inventory (BPI) pain interference scores: Participants rate how much pain interfered with various daily activities, including general activity, walking, work, mood, enjoyment of life, relations with others, and sleep. The interference items is presented with 0-10 scales, with 0=no interference and 10=interferes completely.
Any pain medication or treatment received for relieving pain. If so, the amount of pain relieved. | 3 and 6 months after elective caesarean section
  Currently use of pain medications, its dosages or any other treatment will be recorded.In the last 24 hours, how much relief have pain treatment or medications provided. Please rate in 0-100% where 0% is no relief, 100% complete relief.
Numerical rating Scale (NRS) pain scores and opioid consumption post operatively | 24 and 48 hrs after surgery
  Post operative pain intensity will be assessed using Numerical rating scale(NRS), where 0="no pain" or and 10=pain "as bad as you can imagine." Total opioid consumption will be calculated as total morphine or equivalent in mg.

CONTACTS AND LOCATIONS:
Locations (1):
- BP Koirala Institute of Health Sciences (BPKIHS), Dharān, Koshi, Nepal

IPD SHARING:
Plan to Share IPD: Yes
The final research data will be stored in Mendeley. The final data will be released and shared during the publication process of the manuscript.
Supporting Information: Study Protocol
Time Frame: The final research data and study protocol will be shared with the journal accepting the article for publication. It will be available simultaneously after publication of the article.
Access Criteria: The IPD may be accessed from the link provided in the published manuscript The IPD may also be shared to other researchers by the investigators upon request
URL: https://data.mendeley.com/

REFERENCES:
- [Derived] Subedi A, Schyns-van den Berg AMJV, Thapa P, Limbu PM, Trikhatri Y, Poudel A, Dhakal Y, Bhandari S. Intrathecal morphine does not prevent chronic postsurgical pain after elective Caesarean delivery: a randomised controlled trial. Br J Anaesth. 2022 Apr;128(4):700-707. doi: 10.1016/j.bja.2021.11.036. Epub 2022 Jan 26. PMID 35090722